CLINICAL TRIAL: NCT05976269
Title: The Effects of Bilateral Knee Pain & Dry Needling on Laterality Recognition, Movement, & Function
Brief Title: Bilateral Knee Pain and Dry Needling
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Matt Briggs, Assistant Professor-Practice, Ohio State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020H0332
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Patellofemoral Pain
Keywords: Knee; Dry needling; Acupuncture; Implicit Motor Imagery; Graded Motor Imagery
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Bilateral Patellofemoral Pain with Fear of Movement (Experimental): The first group will consist of 20 subjects presenting with bilateral chronic anterior knee pain and high fear of movement with scores on Tampa Kinesiophobia Scale (fear of movement) greater than 37.
  Interventions: Device: Dry needling
- Bilateral Patellofemoral Pain with Low Fear of Movement (Experimental): The second group with consist of 20 subjects with bilateral chronic anterior knee pain and low fear of movement between ages of 18 and 40 years old.
  Interventions: Device: Dry needling
- Healthy controls without knee pain (Active Comparator): The third group will consist of healthy controls without knee pain between 18 and 40 years old.
  Interventions: Device: Dry needling

INTERVENTIONS:
Device: Dry needling — Dry needling will be performed by licensed physical therapists who are formally trained in dry needling and meet all of the requirements of the state of Ohio and agree to participate as key personnel in this study. These therapists will receive specialized training in the study protocol including appropriate documentation, standardized dry needling technique/procedures, and study communication. Dry needling will be performed in a clean field using sterile acupuncture needles of appropriate length to pierce muscle bellies based on patient size and muscle mass.

SUMMARY:
This project will evaluate the effects of bilateral knee pain and dry needling (DN) on laterality recognition, movement and muscle function. The objective is to determine if laterality recognition accuracy deficits are present in individuals with bilateral chronic knee pain and if DN affects 'central' and 'peripheral' musculoskeletal measurements. Chronic musculoskeletal pain results in changes to the way the brain perceives pain and left-right discrimination between body parts. This phenomenon has been established for individuals with chronic back pain and chronic regional pain syndrome, but has not been described for individuals with bilateral knee pain without the presence of knee OA. Dry needling involves the insertion of a small diameter monofilament needle into muscle, and has been purported to affect the neuromuscular system both centrally and peripherally. Sixty individuals between 18 and 40 years old will be recruited and allocated into three groups. The first group will consist of 20 subjects presenting with bilateral chronic anterior knee pain and high fear of movement with scores on Tampa Kinesiophobia Scale (fear of movement) greater than 37. The second group with consist of 20 subjects with bilateral chronic anterior knee pain and low fear of movement between ages of 18 and 40 years old, and the third group will consist of healthy controls without knee pain between 18 and 40 years old. All subjects will undergo baseline testing consisting of laterality recognition, movement analysis, muscle force production, and ultrasound imaging. Subjects will undergo laterality recognition testing using the Neuro Orthopaedic Institute (NOI) Recognise Knee phone application. 2D video analysis of the lateral step down test will be performed followed by peak isometric force production assessment of knee extension and flexion. Muscle function of the vastus medialis will be measured with ultrasound imaging where cross-sectional area and other measurements (tendon length, muscle thickness, etc) will be captured with Lumify ultrasound imaging transducer. Then DN to the quadriceps will be performed. After DN procedure, subjects will undergo aforementioned measurements from baseline testing. Testing will require only one appointment by the subject, which will last approximately 2 hours an include baseline testing, dry needling, and post testing. No follow up will occur afterwards.

DETAILED DESCRIPTION:
The primary purpose of this study is to identify if a loss of laterality recognition is present in individuals with bilateral chronic knee pain with kinesiophobia and if DN affects short term central and peripheral neuromuscular measurements. The goal of this project is to recruit 20 individuals with bilateral knee pain greater than three months between the ages of 18 and 40 years old without evidence of knee OA and with fear of movement as evidenced by the Tampa Scale of Kinesiophobia with the following aims: Determine if these individuals have a loss of laterality recognition associated with chronic pain that affects the way the brain processes images of a left or right knee using the Neuro Orthopaedic Institute (NOI) Recogonise Knee phone application for iPhone or Android. Assess muscle force production by measuring peak knee extension and flexion isometric force production on a Biodex System II dynamometer (Biodex Medical Systems, Inc. Shirley, New York, USA). Measure muscle function of the quadriceps using ultrasound imaging to assess for changes in cross sectional area, tendon length, muscle thickness, and other relevant measurements that could be captured (i.e. pennation angle) of the vastus medialis (VM) muscle. Assess movement quality with the lateral step down test and using 2D video analysis measure trunk flexion, knee flexion, closed chain dorsiflexion, pelvic drop and patellar projection angle. Determine if DN causes an immediate change on the central (laterality recognition) and peripheral (muscle force production, function, movement) neuromuscular system. Elucidate if there are differences between individuals with bilateral knee pain and high fear of movement and bilateral knee pain and low fear of movement. The investigators also will recruit 20 subjects with bilateral knee pain and low fear of movement, and 20 subjects who are healthy without any knee pain. To the authors knowledge only one study has identified laterality recognition deficits in a population with knee OA. Currently there is not a single publication that assesses laterality recognition deficits for individuals with bilateral knee pain without the presence of knee OA. This study has the potential to inform physical therapists that deliver interventions such as pain neuroscience education, graded motor imagery (left-right discrimination, explicit motor imagery, mirror therapy), movement/muscle function assessment, and DN, to improve their decision-making, evaluation, and treatment skills.

To facilitate recruitment the investigators are applying for a partial HIPAA waiver for this project in order to recruit patients undergoing/seeking care for their knee pain with a physician or physical therapist. The only pertinent PHI to be screened will be age, diagnosis codes related to knee pain, and factors related to inclusion and exclusion criteria. Of this information, only eligibility criteria (inclusion/exclusion factors) will be screened by the research team. This information screened in the electronic medical record will not be written down or stored anywhere. Once a research associate identifies a patient that may qualify for the study, the patient will fill out a survey link from REDCap, where the data will be stored containing their name, contact information, and screening questions related to their eligibility of the study (inclusion/exclusion criteria). This information will be preserved in REDCap, a secure online platform for data storage, for the sole purpose of avoiding contacting subjects repetitively regarding interest in study participation. Only pertinent PHI will be screened such as age, diagnosis codes related to knee pain, and factors related to inclusion and exclusion criteria. None of this information will be stored by the research team. Once a research associate identifies a patient that may qualify for the study, the patient will fill out a survey link from REDCap, where the data will be stored containing their name, contact information, and screening questions related to their eligibility of the study. Participants in this study do not have to be current patients. If a potential participant who is not a current patient reaches out to the research team, they will be given the survey link from REDCap. After this survey is completed, a research associate will determine their eligibility for the study. This means recruits for the study may come from the community who have not necessarily seen a PT, MD, or DO. All interventions, including dry needling, and outcomes measured (pain, outcome questionnaires, strength, range of motion, functional assessment, etc.) are commonly performed during current physical therapy practice and treatment. For this study the investigators are formalizing the collection of these measures. Testing will require only one appointment by the subject, which will last approximately 2 hours an include baseline testing, dry needling, and post testing. No follow up will occur afterwards. Specific testing procedures related to this protocol include the following: Laterality recognition testing, where the subject will look through an application called NOI Recognoise Knee on an iPhone or iPad and select if the image they are looking at is a left or right knee. Cross-sectional area and other measurements (tendon length, muscle thickness, etc) of vastus medialis muscle measured in supine with Lumify ultrasound imaging transducer. 2D movement analysis will be performed of subjects performing the lateral step down test. Peak knee extension and flexion isometric force production will be captured using the Biodex. Dry needling will be provided to all subjects using a clean technique commonly used in clinical care. Dry needling intervention will be provided to the quadriceps muscle using a standardized protocol. Dry needle will be inserted in and out and/or twisted clockwise for a maximum of 30" at the discretion of the researcher and tolerance of participant, and then the needle will be left in situ for 15 minutes. Several studies have demonstrated the safety of this technique. If participant is unable to tolerate the DN procedure, the procedure will be stopped and needles removed. The participant can stop participation at any time during the study. Step 1-4 will be repeated. In summary, the process will look like this: Consent, Baseline testing, dry needling, post testing in a 2 hour session. In addition, specific examination data from the subjects' will be recorded such as age, height, weight and details about their knee pain. Both electronic and paper collection of data and questionnaires will be used for the study. This study will utilize REDCap (Research Electronic Data Capture), a software tool set and workflow methodology for electronic collection and management of clinical and research data, to collect and store data. REDCap will be used as the primary tool to collect and manage the study documentation as it pertains to the screening, data collection, and participant questionnaires. Paper documentation will also be available. The paper documentation would be used if the REDCap system could not be accessible for some reason including but not limited to internet outage, computer technical difficulties (hardware and/or software), loss of power, etc.

Testing will require only one appointment by the subject, which will last approximately 2 hours an include baseline testing, dry needling, and post testing. No follow up will occur afterwards. Once subjects have been screened and have agreed to be included in the study they will be scheduled for a 2 hour testing session. The subject will then undergo informed consent, baseline testing, dry needling, and post testing. Currently the investigators only have funding for 10 subjects who have bilateral knee pain and high fear of movement. They will receive a consent form that details the honorarium they will receive. Those who meet the inclusion criteria of the other groups that investigators don't have funding for, will receive a different consent and hippa form that has all the same details as the other form without the honorarium information. Testing will take approximately 2 hours. 10 minutes will be allocated for consent and questions. 45 minutes will be allocated to the baseline testing. 15 minutes will be allocated to the dry needling procedure. 45 minutes will be allocated for post testing. 5 minutes will be allocated for concluding the study. Summary of two hour testing session Step 1: Consent Subject: subjects will have already filled out screening questionnaire (inclusions criteria Table 1). The informed consent process will occur and patients will be given the option to consent to participate and continue in the study. Step 2: Laterality Recognition: Basic - Images of left and right knees with plain background Vanilla - Basic images of left and right knees in different orientations Context - Images of left and right knees in real life activities Abstract - Images of left and right knees with various artwork and statues Step 3: Lateral Step Down Test: 2D video analysis performed with two Go Pros to capture the five repetitions of subject performing lateral step down test in frontal and sagittal plane. Step 4: Muscle Force Production: Peak knee extension and flexion isometric force production captured on Biodex. Step 5: Muscle Function: Cross-sectional area of vastus medialis muscle measured in supine with Lumify ultrasound imaging transducer. Step 6: Dry Needling: Dry needles inserted into distal vastus lateralis, rectus femoris and vastus medialis muscles. Needle inserted maximally and left in situ for 15 minutes. Step 7: Repeat steps 2 thru 5: Repeat laterality recognition testing, lateral step down test, muscle force production, and muscle function testing.

The investigators plan to recruit 60 subjects; 40 with bilateral knee pain and divide them in two different groups: high fear (Tampa Kinesiophobia Scale > 37), low fear (Tampa Kinesiophobia Scale = or < 37), and 20 healthy controls into a group without knee pain. In order to be adequately powered, our goal is to recruit 20 subjects per group. Currently the investigators only have funding for 10 subjects who have bilateral knee pain and high fear of movement. They will receive a consent form that details the honorarium they will receive. Those who meet the inclusion criteria of the other groups that investigators don't have funding for, will receive a different consent and hippa form that has all the same details as the other form without the honorarium information. Based on previous research and sample size power calculation using the statistical analysis software STATA, 10 subjects are required to yield a medium effect size, alpha level of 0.01 and power level of 0.80. This meets our goal of being adequately powered to assess for laterality recognition deficits, however the investigators plan to recruit 60 total subjects with 20 subjects for each group so the investigators can be adequately powered to assess for differences in each group for all mentioned variables.

ELIGIBILITY:
Inclusion Criteria:

* For high fear group: Age between 18 and 40 years old, pain greater than or equal to 3 months, Tampa scale of kinesiophobia >37, anterior knee pain scale <90, and no evidence of knee OA
* For low fear group: Age between 18 and 40 years old, pain greater than or equal to 3 months, Tampa scale of kinesiophobia <37, anterior knee pain scale <90, and no evidence of knee OA
* For control group: no surgery in past 6 months, age between 18 and 40 years old, no knee OA, Tampa Scale <10, and anterior knee pains scale >90

Exclusion Criteria:

* Knee surgery in past 6 months, previous dry needling or acupuncture to knee, pregnancy, menicscal/cartilage/ligamentous injury, history of patellar subluxations, dislocations, or MPFL reconstruction, contraindications to dry needling or acupuncture, or neurological condition that affects movement.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2028-07-21 (Estimated); Study Completion 2030-07-21 (Estimated)

PRIMARY OUTCOMES:
Accuracy and response time from left right judgement task | Complete immediately before, and immediately after dry needling procedure.
  This is referred to as implicit motor imagery performance and participants have to accurately identify if a group of randomized knee images is a left or a right.

SECONDARY OUTCOMES:
2D Video Assessment of Movement Patterns During Lateral step down test. | Complete immediately before, and immediately after dry needling procedure.
  Participant will perform lateral step down test while GoPro videos capture the movement.
Muscle depth of of vastus medialis oblique muscle as measured by Lumify US unit | Complete immediately before and immediately after dry needling procedure.
  Depth of muscle will be measured with diagnostic US.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Briggs, DPT, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Jameson Crane Sports Medicine Institute, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No